CLINICAL TRIAL: NCT01606800
Title: Randomized Open Label Study to Assess the Efficacy and Safety of Short Course Therapy (24 Weeks) With Peginterferon Alpha-2b and Ribavirin for Chronic Hepatitis C (Genotype 4) Patients Who Achieve a Rapid Virological Response (HCV -RNA Undetectable at Week 4 of Treatment)
Brief Title: Efficacy and Safety of Short Course Therapy With Peginterferon Alpha-2b (PEG-IFN Alfa-2b) and Ribavirin (RBV) for Chronic Hepatitis C (Genotype 4) Participants Achieving a Rapid Virological Response at Week 4 of Treatment (MK-8908B-059)
Acronym: START 4
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The trial was terminated due to change in new standard of therapy during the study period.
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8908B-059; MK-8908B-059 (Other: Merck Registration Number)
Record Dates: First submitted 2012-05-24; First posted 2012-05-28 (Estimated); Results first posted 2016-02-23 (Estimated); Last update posted 2018-10-25 (Actual); Status verified 2018-09

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 44 Weeks of PEG-IFN alfa-2b + RBV (Experimental): Participants achieving RVR at 4 weeks of treatment will receive 44 additional weeks of Peg-IFN Alfa-2b + RBV.
  Interventions: Drug: PEG-IFN alfa-2b; Drug: ribavirin
- 20 Weeks of PEG-IFN alfa-2b + RBV (Experimental): Participants achieving RVR at 4 weeks of treatment will receive 20 additional weeks of Peg-IFN Alfa-2b + RBV.
  Interventions: Drug: PEG-IFN alfa-2b; Drug: ribavirin

INTERVENTIONS:
Drug: PEG-IFN alfa-2b — Pegylated interferon alfa-2b administered subcutaneously 1.5 mcg/kg/week
Drug: ribavirin — Ribavirin 200 mg capsules administered orally daily based on weight

SUMMARY:
The purpose of this study is to assess the efficacy of a short course of therapy (24 weeks) versus standard 48 week treatment in previously untreated adult participants with chronic hepatitis C (CHC) genotype 4 infection who achieve rapid virologic response (RVR), defined as HCV ribonucleic acid (RNA) negativity after 4 weeks of treatment.

DETAILED DESCRIPTION:
Participants who achieved RVR after 4 weeks of PEG-INF alfa-2b plus RBV treatment were randomized to receive either 20 or 44 weeks of continued therapy, for a total of 24 or 48 weeks total of PEG-INF plus RBV therapy.

ELIGIBILITY:
Inclusion Criteria:

* Participant is ≥40 kg and ≤120 kg weight
* Participant and participant's partner(s) must each agree to use acceptable methods of contraception for at least 2 weeks prior to Day 1 and continue until at least 6 months after last dose of study medication, or longer if dictated by local regulations.
* Previously documented CHC genotype 4 infection
* Liver biopsy or fibrotest and fibroscan with histology consistent with CHC and no other etiology and with hepatic fibrosis scores (F0, F1, F2, F3).

Exclusion Criteria:

* Co-infected with the human immunodeficiency virus (HIV) or hepatitis B virus
* Treatment for hepatitis C with any investigational medication
* Treatment with any investigational drug within 30 days of the screening visit
* Evidence of decompensated liver disease including, but not limited to, a history or presence of clinical ascites, bleeding varices, or hepatic encephalopathy
* Autoimmune hepatitis or a history of autoimmune disease
* Hepatic fibrosis score F4
* Severe pre-existing cardiac disease, including unstable or uncontrolled cardiac disease in the previous six months
* Autoimmune hepatitis or a history of autoimmune disease
* Thyroid disease uncontrolled with conventional treatment
* Epilepsy and/or compromised central nervous system (CNS) function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2015-01-26 (Actual); Study Completion 2015-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=8908B-059&kw=8908B-059&tab=access

RESULTS

PARTICIPANT FLOW:
Groups:
- 44 Weeks of PEG-IFN Alfa-2b + RBV: Participants achieving rapid virologic response (RVR) after 4 weeks of pegylated interferon (PEG-INF) alfa-2b + ribavirin (RBV) treatment continued to receive PEG-INF alpha-2b + RBV for an additional 44 weeks.
- 20 Weeks of PEG-IFN Alfa-2b + RBV: Participants achieving RVR after 4 weeks of PEG-INF alfa-2b + RBV treatment continued to receive PEG-INF alpha-2b + RBV for an additional 20 weeks.
Period: Overall Study
Arm/Group | 44 Weeks of PEG-IFN Alfa-2b + RBV | 20 Weeks of PEG-IFN Alfa-2b + RBV
Started | 22 | 23
Treated | 22 | 23
Completed | 17 | 21
Not Completed | 5 | 2
Not completed — Adverse Event | 3 | 1
Not completed — Participant withdrew consent | 0 | 1
Not completed — Missing completion status | 2 | 0

BASELINE CHARACTERISTICS:
Population: All Treated Population, which included all participants who received at least one dose of study medication after RVR.
Groups:
- Total: Total of all reporting groups
Arm/Group | 44 Weeks of PEG-IFN Alfa-2b + RBV | 20 Weeks of PEG-IFN Alfa-2b + RBV | Total
Number analyzed (Participants) | 22 | 23 | 45
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.4 (10.79) | 37.1 (11.22) | 37.7 (10.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 13 | 13 | 26

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Achieving Sustained Virologic Response (SVR)
Description: SVR was defined as undetectable HCV RNA levels 24 weeks after the completion of therapy.
Time Frame: At 24 weeks after the completion of therapy (up to 72 weeks)
Population: All Treated Population, which included all participants who received at least one dose of study medication after RVR.
Measure: Number; unit: Participants
Arm/Group | 44 Weeks of PEG-IFN Alfa-2b + RBV | 20 Weeks of PEG-IFN Alfa-2b + RBV
Number analyzed (Participants) | 22 | 23
Participants | 13 | 22

ADVERSE EVENTS:
Time Frame: Up to 72 weeks
Description: All Treated Population, which included all participants who received at least one dose of study medication after RVR.
Arm/Group | 44 Weeks of PEG-IFN Alfa-2b + RBV | 20 Weeks of PEG-IFN Alfa-2b + RBV
Serious Adverse Events (participants affected / at risk) | 0/22 | 2/23
Other Adverse Events (participants affected / at risk) | 16/22 | 13/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 44 Weeks of PEG-IFN Alfa-2b + RBV (N=22) | 20 Weeks of PEG-IFN Alfa-2b + RBV (N=23)
Anemia (Blood and lymphatic system disorders) | 0 | 1
Leukopaenia (Blood and lymphatic system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 44 Weeks of PEG-IFN Alfa-2b + RBV (N=22) | 20 Weeks of PEG-IFN Alfa-2b + RBV (N=23)
Anemia (Blood and lymphatic system disorders) | 5 | 2
Vision blurred (Eye disorders) | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1
Fatigue (General disorders) | 5 | 1
Pyrexia (General disorders) | 2 | 0
Blood thyroid stimulating hormone increased (Investigations) | 2 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Headache (Nervous system disorders) | 3 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2

LIMITATIONS AND CAVEATS:
This Trial was prematurely terminated due to the availability of more promising treatment for HCV participants and the change in treatment guidelines, which will offer the patient a better treatment opportunity.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to provide to the sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication (including, without limitation, slides and texts of oral or other public presentations and texts of any transmission through any electronic media, eg, any computer access system such as the Internet, World Wide Web, etc) that report any results of the trial.